CLINICAL TRIAL: NCT06326047
Title: Investigation of the Safety and Efficacy of Once Weekly NNC0519-0130 in Participants With Type 2 Diabetes - a Dose Finding Study
Brief Title: A Research Study Comparing How Well Different Doses of the Medicine NN0519-0130 Lower Blood Sugar in People With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9541-4945; U1111-1291-9196 (Other: World Health Organization (WHO)); jRCT2031230704 (Registry Identifier: JRCT)
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures. The study will be double-blinded within dose level of once weekly subcutaneously administered NNC0519-0130 and the corresponding volume-matched placebo arms. The active comparator arm with tirzepatide will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Dosing scheme A (NNC0519-0130) (Experimental): Participants will receive NNC0519-0130 at 3 dose levels once weekly (QW) as subcutaneous (s.c.) injection in dose escalating manner.
  Interventions: Drug: NNC0519-0130
- Dosing scheme A (Placebo) (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo once weekly s.c. for 3 periods.
  Interventions: Drug: Placebo
- Dosing scheme B (NNC0519-0130) (Experimental): Participants will receive NNC0519-0130 at 3 dose levels once weekly (QW) as s.c. injection in dose escalating manner.
  Interventions: Drug: NNC0519-0130
- Dosing scheme B (Placebo) (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo once weekly s.c. for 3 periods.
  Interventions: Drug: Placebo
- Dosing scheme C (NNC0519-0130) (Experimental): Participants will receive NNC0519-0130 at 5 dose levels once weekly as s.c. injection in dose escalating manner.
  Interventions: Drug: NNC0519-0130
- Dosing scheme C (Placebo) (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo once weekly s.c. for 3 periods.
  Interventions: Drug: Placebo
- Dosing scheme D (NNC0519-0130) (Experimental): Participants will receive NNC0519-0130 at 5 dose levels once weekly as s.c. injection in dose escalating manner.
  Interventions: Drug: NNC0519-0130
- Dosing scheme D (Placebo) (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo once weekly s.c. for 3 periods.
  Interventions: Drug: Placebo
- Dosing scheme E (NNC0519-0130) (Experimental): Participants will receive NNC0519-0130 at 7 dose levels once weekly as s.c. injection in dose escalating manner.
  Interventions: Drug: NNC0519-0130
- Dosing scheme E (Placebo) (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo once weekly s.c. for 3 periods.
  Interventions: Drug: Placebo
- Dosing scheme F (tirzepatide) (Active Comparator): Participants will receive tirzepatide at 6 dose levels once weekly as s.c. injection in dose escalating manner.
  Interventions: Drug: Trizepatide

INTERVENTIONS:
Drug: NNC0519-0130 — NNC0519-0130 will be administered subcutaneously.
  Arms: Dosing scheme A (NNC0519-0130); Dosing scheme B (NNC0519-0130); Dosing scheme C (NNC0519-0130); Dosing scheme D (NNC0519-0130); Dosing scheme E (NNC0519-0130)
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Dosing scheme A (Placebo); Dosing scheme B (Placebo); Dosing scheme C (Placebo); Dosing scheme D (Placebo); Dosing scheme E (Placebo)
Drug: Trizepatide — Trizepatide will be administered subcutaneously.
  Arms: Dosing scheme F (tirzepatide)

SUMMARY:
This study will look at how well a new medicine called NNC0519-0130 helps people with type 2 diabetes lower their blood sugar and body weight. The study will test up to 7 different doses of NNC0519-0130. Which treatment participant will get is decided by chance. Participants will take 1-3 injections once a week. The study medicine will be injected under skin with a thin needle in the stomach, thigh, or upper arm. The study will last for about 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential, or male.
* For United States (US) only: Female of childbearing potential using highly effective non-systemic methods of contraception with low user-dependency and willingness to continue using it through-out the study or male.
* Age 18-75 years (both inclusive) at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus greater than or equal 180 days before screening.
* Stable daily dose(s) more than or equal 90 days before screening of the following antidiabetic drug(s) or combination regimen(s) at effective or maximum tolerated dose as judged by the investigator: metformin with or without sodium-glucose co-transporter 2 (SGLT2) inhibitor.
* Glycated haemoglobin (HbA1c) of 7.5-10.0% (58-86 millimoles per moles (mmol/mol)) (both inclusive) as assessed by central laboratory at screening.
* Body mass index (BMI) greater than or equal 23.0 kilograms per meter square (kg/m^2).

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 consecutive days and prior insulin treatment for gestational diabetes are allowed.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire question.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Change in Glycated haemoglobin (HbA1c) | From baseline (week 0) to 12 weeks on a given maintenance dose
  Measured as percentage point (%-point)

SECONDARY OUTCOMES:
Change in Glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 36)
  Measured as percentage point (%-point)
Relative change in body weight | From baseline (week 0) to end of treatment (week 36)
  Measured as percentage (%)
Change in body weight | From baseline (week 0) to end of treatment (week 36)
  Measured as kilograms (kg)
Change in fasting plasma glucose (FPG) | From baseline (week 0) to 12 weeks on a given maintenance dose
  Measured as millimoles per liter (mmol/L)
Continuous glucose monitoring (CGM): Change in time in range (TIR) 3.9-10.0 millimoles per liter (mmol/L) (70-180 milligrams per deciliter (mg/dL)) | From baseline (week -2 to week 0) to week 22-24 and week 34-36, respectively
  Measured as percentage point (%-point)
Change in waist circumference | From baseline (week 0) to end of treatment (week 36)
  Measured as centimeter (cm)
Change in systolic blood pressure (SBP) | From baseline (week 0) to end of treatment (week 36)
  Measured as millimeters of mercury (mmHg)
Change in high sensitivity C-Reactive Protein (hsCRP) | From baseline (week 0) to end of treatment (week 36)
  Measured as ratio to baseline
Change in total cholesterol | From baseline (week 0) to end of treatment (week 36)
  Measured as ratio to baseline
Change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 36)
  Measured as ratio to baseline
Change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 36)
  Measured as ratio to baseline
Change in triglycerides | From baseline (week 0) to end of treatment (week 36)
  Measured as ratio to baseline
Number of adverse events | From baseline (week 0) to end of study (week 40)
  Measured as number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (94):
- United States (49):
  - Velocity Clin Res-Chula Vista, Chula Vista, California
  - Valley Research, Fresno, California
  - 310 Clinical Research, Inglewood, California
  - Velocity Clin Res San Diego, La Mesa, California
  - First Valley Med Grp Lancaster, Lancaster, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Catalina Research Institute, LLC, Montclair, California
  - Med Partners, Inc., Toluca Lake, California
  - UCLA Health Southbay Endocrine, Torrance, California
  - University Clin Investigators, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - Innovative Research of W Florida Inc., Clearwater, Florida
  - Innovative Research of W FL, Clearwater, Florida
  - International Research Associates, LLC_Miami, Miami, Florida
  - Centricity Research, Columbus, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Centennial Medical Group, Columbia, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Endo And Metab Cons, Rockville, Maryland
  - Clinvest Research, Springfield, Missouri
  - Mercury Str Med Grp, PLLC, Butte, Montana
  - Excel Clinical Network, Las Vegas, Nevada
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Velocity Clinical Research Binghamton, Binghamton, New York
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare Wilmington, Wilmington, North Carolina
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Velocity Clin Res_Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research Springdale, Cincinnati, Ohio
  - Providence Health Partners Ctr, Dayton, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - Tristar Clin Investigations, PC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians Inc., Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Uniontown, Pennsylvania
  - Velocity Clinical Research Abilene, Abilene, Texas
  - Tekton Research, Austin, Texas
  - Velocity Clin Res Austin, Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Zenos Clinical research, Dallas, Texas
  - Care United Research, LLC, Forney, Texas
  - Endocrine Associates Houston, Houston, Texas
  - Biopharma Informatic_Houston, Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Burke Internal Medicine & Research, Burke, Virginia
  - TPMG Clinical Research, Newport News, Virginia
- Australia (10):
  - Macquarie University, Macquarie Park, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Roger Chih Yu Chen, Sydney, New South Wales
  - Western Endocrine Blacktown, Sydney, New South Wales
  - Illawarra Diabetes Service Clinical Trials & Research Unit, Wollongong, New South Wales
  - University of Sunshine Coast, Birtinya, Queensland
  - Eastern Clinical Research Unit Box Hill, Box Hill, Victoria
  - Emeritus Research Melbourne, Camberwell, Victoria
  - Austin Health, Metabolic Disorders Centre, Heidelberg Heights, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Canada (11):
  - OCT Research ULC (dba Okanagan Clinical Trials), Kelowna, British Columbia
  - OCT Research ULC (dba Okanagan Clinical Trials), Richmond, British Columbia
  - Cook Street Medical Clinic, Victoria, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Albion Finch Medical Centre, Toronto, Ontario
  - Centricity Research Quebec City, Lévis, Quebec
  - Recherche GCP Research, Montreal, Quebec
  - Centricity Research Ville St. Laurent VSL, Saint-Laurent, Quebec
  - Diex Recherche Quebec Inc., Québec
- India (9):
  - Life Care Hospital and Research Centre, Bangalore, Karnataka
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - Diabetes Research Center, Hyderabad, Hyderabad, Telangana
  - MS Ramaiah, Bengaluru
- Japan (5):
  - Tokuyama clinic_Diabetic internal medicine, Chiba
  - Soka Sugiura Internal Medicine Clinic, Soka-shi, Saitama
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic, Tokyo
- South Africa (5):
  - Josha Research, Bloemfontein, Free State
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Shop#1 Health Emporium, Midrand, Gauteng
  - Dr Pillay's Rooms, Durban, KwaZulu-Natal
  - Dr T Padayachee, eMkhomazi, KwaZulu-Natal
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com